CLINICAL TRIAL: NCT02694783
Title: A Pilot Study of Adoptive Cellular Immunotherapy for Progressive Multifocal Leukoencephalopathy With Ex Vivo Generated Polyomavirus-Specific T-cells
Brief Title: Adoptive Cellular Immunotherapy for Progressive Multifocal Leukoencephalopathy With Ex Vivo Generated Polyomavirus-Specific T-Cells
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160072; 16-N-0072
Record Dates: First submitted 2016-02-27; First posted 2016-03-01 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-06-10

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: HLA Matched; JCV; Donor; PyVST; PML
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): ex vivo generated polyomavirus-specific T cells from HLA-matched donor
  Interventions: Biological: PyVST

INTERVENTIONS:
Biological: PyVST — ex vivo generated polyomavirus-specific T cells from HLA-matched donor

SUMMARY:
Background:

Progressive Multifocal Leukoencephalopathy (PML) is a brain infection in people with a weakened immune system. Researchers think polyoma virus specific T cells (PyVST) therapy can treat PML. The PyVST cells are made from blood cells of a healthy relative. They are grown in a lab to expand the virus-killing cells, then given to the person with PML.

Objective:

To test whether PyVST safely treats PML.

Eligibility:

* Adults ages 18 and older with PML
* Healthy adults ages 18 and older who have:

  * Been screened under protocol 97-H-0041
  * A sibling, parent, or child with PML and matching cells

Design:

* Participants will be screened with:

  * Medical history
  * Physical exam
  * Blood and urine tests
* PML participants will also be screened with:

  * Cerebrospinal fluid removed by needle in the back.
  * MRI: A dye is injected in a vein. They lie on a table that slides into a cylinder.
  * Questionnaires

Healthy participants will have apheresis: Blood flows through a needle in one arm into machine that separates blood cells needed for donation. The rest of the blood is returned by needle to the other arm. Some participants may have a central line placed in a vein instead. They can have apheresis up to 3 times, at least 28 days apart.

Participants with PML will receive the PyVST cells by needle in the arm. They will stay in the hospital 1 week. They can do this up to 3 times, at least 28 days apart. After each infusion, they will have weekly visits for 1 month. Then they will have 4 visits over 1 year. Visits include repeats of screening tests.

DETAILED DESCRIPTION:
Objective

This pilot clinical trial will aim to determine the feasibility and potential toxicities associated with treating patients with progressive multifocal leukoencephalopathy (PML) with polyomavirus (PyV)-specific partially matched polyclonal allogeneic T cells. It will further provide initial efficacy data for this indication.

Study Population

Up to 18 subjects with definite PML, defined as clinical signs and MRI compatible with active PML and the presence of JCV by PCR in CSF. Subjects must be 18 years of age or older and must have a first degree, partially HLA- matched relative able and willing to act as a donor of lymphocytes. Subjects with underlying reversible immunosuppression (i.e.- HIV or MS status post treatment with natalizumab), or subjects with uncontrolled malignancy will be excluded. Subjects with evidence of active CNS inflammation as determined by presence of significant contrast enhancement within the PML lesions by MRI will also be excluded because it is assumed such patients are already mounting an adequate immune response against the infection.

Design

This will be a first-in-human pilot study assessing the feasibility and toxicity profile of NIH PyVST cellular product in subjects with PML. Subjects will be screened under the existing NIH Natural History study of PML (13-N-0017). Sequential enrollment will be spaced at least 28 days apart. An initial fixed dose PyVST infusion (target dose of 1 x 10(6) PyVST/kg (+/- 10%)) will be administered by intravenous (IV) infusion, followed by 2x 10(6) PyVST/kg (+/-10%) up to 2 times to each subject if needed.

Outcome Measures

Safety will be monitored to 28 days continuously with stopping rules based on the treatment-related serious adverse event rate. Secondary outcomes include survival, assessed at day 28 and at 1 year following the last infusion. CSF viral titers, MR imaging, and clinical disability scales will also be collected.

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENT:
* Clinically definite PML, defined as clinical signs and MRI compatible with active PML and the presence of JCV by PCR in CSF
* Modified Rankin Scale 1-4, inclusive
* Age 18 or older
* Patient medically stable and able to tolerate travel to NIH
* Available PyVST
* Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study
* Willing and able to participate in all aspects of trial design and follow-up
* Able to provide informed consent at the time of study enrollment (not required for reinfusions).

EXCLUSION CRITERIA - PATIENT:

* Patients with human immunodeficiency virus (HIV infection)
* Patients who have been treated with natalizumab
* Patients with readily reversible immunosuppressive state
* Patients receiving immunosuppressive or immunomodulatory therapies within 28 days of screening for enrollment that could interfere with PyVST function
* Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections, patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.
* Patients who have received donor lymphocyte infusion (DLI) within 28 days
* Uncontrolled relapse of malignancy
* Patients with any other associated CNS disease that might confound outcomes
* Patients with contraindication to MRI (including cardiac pacemakers and some infusion pumps, other metallic implants, metallic foreign objects)
* MRI findings consistent with immune system reconstitution inflammatory syndrome (IRIS) and determined to be mounting an adequate immune response to the infection
* Patients with medical contraindication to LP
* For subjects who have previously received PyVST infusions, any treatment-limiting toxicity (defined in Section 8.3) to previous infusions
* Subjects with a positive pregnancy test or who are nursing.

INCLUSION CRITERIA - DONOR:

* Ability to provide informed consent at the time of enrollment
* First degree relative of patient (sibling, parent/child)
* Age 18 or older

EXCLUSION CRITERIA - DONOR:

* Sickling hemoglobinopathies including HbSS and HbSC by history and peripheral blood smear; donors with HbAS are acceptable
* HbsAg, anti-HBc, anti-HCV, anti-HIV, anti-HTLV, and RPR
* Cardiovascular instability, severe anemia, inadequate venous access, severe coagulation disorder or any other medical condition that the Principal Investigator or Apheresis Unit staff considers a contraindication to the apheresis procedure or research blood draw.
* Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Characterization of the safety and feasibility of PyVST infusion for the treatment of PML based on development of Treatment Limiting Toxicity | ongoing
  Characterization of the safety and feasibility of PyVST infusion for the treatment of PML based on development of Treatment Limiting Toxicity

SECONDARY OUTCOMES:
PML lesion volume | change from baseline to day 28
  Change from baseline to day 28 in PML lesion volume, as seen on brain MRI
Gadolinium enhancement | Change in pattern of gadolinium enhancement from baseline to day 3, day 7, day 14, and day 28
  Change in pattern of gadolinium enhancement from baseline to day 3, day 7, day 14, and day 28 MRI scans of participants' brains
Modified Rankin Score | Change from baseline to day 28
  Change from baseline to day 28 in the modified Rankin Score (mRS).
JC viral load in CSF | Change from baseline to day 28
  Change from baseline to day 28 in JC viral load in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Irene CM Cortese, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Cortese I, Beck ES, Al-Louzi O, Ohayon J, Andrada F, Osuorah I, Dwyer J, Billioux BJ, Dargah-Zada N, Schindler MK, Binder K, Reoma L, Norato G, Enose-Akahata Y, Smith BR, Monaco MC, Major EO, Jacobson S, Stroncek D, Highfill S, Panch S, Reich DS, Barrett J, Nath A, Muranski P. BK virus-specific T cells for immunotherapy of progressive multifocal leukoencephalopathy: an open-label, single-cohort pilot study. Lancet Neurol. 2021 Aug;20(8):639-652. doi: 10.1016/S1474-4422(21)00174-5. PMID 34302788
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-N-0072.html